CLINICAL TRIAL: NCT00937222
Title: Effects of Peanut and Peanut Butter Consumption on Blood Lipids and Glycemic Control in Adults Ith Type 2 Diabetes
Brief Title: Effects of Peanut and Peanut Butter Consumption on Blood Lipids and Glycemic Control in Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: National Peanut Board (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, Principal Investigator, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59049
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; cholesterol; peanuts; peanut butter; dietary intervention; HDL cholesterol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Peanuts and peanut butter — Peanuts and peanut butter

SUMMARY:
Peanuts and peanut butter contain high levels of monounsaturated fat (MUFA), arginine, fiber, phytosterols, resveratrol and vitamin E that have the potential to reduce cardiovascular disease (CVD) risk through improved blood glucose control and favorable modification of blood lipids. When substituted for saturated fat in the diet, MUFA may have important metabolic benefits for persons with diabetes. Therefore, the investigators propose to study the effects of a peanut and peanut butter-enriched diet on markers of CVD risk factors in free-living adults with diabetes residing in Southern California. This study's primary clinical outcome will be high-density lipoprotein (HDL) - cholesterol. Secondary outcomes will include additional serum lipids (total cholesterol, low-density lipoprotein (LDL) - cholesterol and triacylglycerol), glucose, HbA1c, and anthropometry (body weight, body composition and waist circumference). This study will provide vital information about the role of peanuts and peanut butter in modulating blood glucose homeostasis and CVD risk factors among adults with diabetes.

DETAILED DESCRIPTION:
This will be a parallel randomized controlled intervention study on free-living adults with diabetes. The study duration will be 6 months. Participants will be randomized to receive one of two dietary approaches (moderate fat, control; and, moderate fat inclusive of 32 g peanuts or 2 Tbsp. peanut butter per day, intervention) to an ADA meal plan targeting a profile of 35% fat, 45% CHO and 20% protein. A supply of peanuts and peanut butter from the National Peanut Board will be provided to participants assigned to the intervention group at clinic visits. The peanuts and peanut butter will be consumed as part of the participant's customary meals and snacks. In light of ADA's prior recommendation to derive 60 to 70% of energy intake from CHO and MUFA, the peanuts and peanut butter will provide an enhanced proportion of energy from MUFA (total fat content of peanuts by compositional weight is 22% and 52% of the total fat is MUFA).

An experienced Registered Dietitian and Certified Diabetes Educator will oversee the dietary advice provided to each of the two groups. All participants will be provided with an individualized portion-controlled meal plan using the ADA food exchange lists and possibly modified fat instruction on fatty acid considerations and inclusion of peanuts and peanut butter. Dietary compliance, especially the intake of peanuts and peanut butter, will be measured by six 24-hour recalls without notice (telephone interview by a dietitian on what was consumed the previous day). Participants will be requested to maintain their activities and other lifestyle habits and to record in diaries provided to them any signs of illness, medications used, and any deviation from their prescribed diet. The investigators will examine diaries at the clinic visits. No major deviations from the protocol will be tolerated.

Less than 100 ml of blood will be drawn from each participant at baseline (week 0), week 12 and week 24. All blood drawings will be performed at Loma Linda University Medical Center. Participants will report to the laboratory on the assigned days after fasting for a minimum of 12 hours. Body weight and body composition measurements (percent body fat, fat free mass, total body water) will be obtained at each clinic visit using an internally calibrated segmental bioelectrical impedance analysis device (Tanita®, Arlington Heights, IL).

ELIGIBILITY:
Inclusion Criteria:

* Presence of a medical diagnosis of diabetes for at least 6 months
* HbA1c < 9%
* Age greater than 18 years
* Resident of Loma Linda, California area

Exclusion Criteria:

* Allergy to peanuts
* Smokers
* History of irritable bowel disease or diverticulitis
* Statin therapy (unless stable statin dose for 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is HDL-C | 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Serum lipids, glucose, HbA1c, anthropometrics and blood pressure | 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabaté, MD, DrPh, Principal Investigator — Chair, Department of Nutrition; Michelle Wien, DrPH, Study Director — Assistant Professor, Department of Nutrition
Locations (1):
- Loma Linda University Medical Center Diabetes Treatment Center, Loma Linda, California, United States

REFERENCES:
- [Derived] Wien M, Oda K, Sabate J. A randomized controlled trial to evaluate the effect of incorporating peanuts into an American Diabetes Association meal plan on the nutrient profile of the total diet and cardiometabolic parameters of adults with type 2 diabetes. Nutr J. 2014 Jan 22;13:10. doi: 10.1186/1475-2891-13-10. PMID 24450471
- See also: Related Info — http://www.nutstudies.org/currentstudies.html